CLINICAL TRIAL: NCT06473532
Title: TEXT4HF: A Randomized Controlled Trial of a Tailored Text Messaging Intervention to Improve Self-Care in Older Adult Patients With Heart Failure
Acronym: TEXT4HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jonathan W. Leigh, PhD Candidate, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0704
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; mHealth; Text Messaging; Mobile Phone
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEXT4HF (Experimental): In addition to usual care and a standard AHA information packet for patients with HF, participants in the intervention group will receive 5 tailored TMs/week for 12 weeks, targeting health beliefs about medication adherence, heart-healthy diet, self-monitoring, and heart failure knowledge.
  Interventions: Behavioral: TEXT4HF
- Control Group (No Intervention): The control group will receive standard HF medical care, which includes nurse-led patient education about HF self-care before and/or after discharge as well as follow-up visits at the Outpatient Heart Failure Clinic at UIH post-hospital discharge and several times per year or more, depending on the severity of the patient's condition. Participants will also receive the AHA information packet for patients with HF.

INTERVENTIONS:
Behavioral: TEXT4HF — In addition to usual care, participants in the intervention group will receive 5 TMs/week for 12 weeks at a time of their preference. Tailoring of the TMs is performed based on participants' responses to validated questionnaires (health beliefs scales, HF-knowledge scale, and self-efficacy about HF self-care scale), administered at baseline and 4 weeks. They will also receive an AHA HF discharge informational packet.
  Arms: TEXT4HF

SUMMARY:
The goal of this study is to determine whether an individually tailored text messaging intervention can improve self-care in older adult patients with heart failure. The main question it aims to answer are:

* Is a tailored text messaging intervention feasible and acceptable among older adult patients with heart failure?
* Does tailored text messaging improve self-care in adult patients with heart failure?

Participants will be randomly assigned to one of two groups for 12 weeks: 1) intervention (text messaging); or 2) control group. Both groups will receive usual care, which includes regular follow-up visits at the heart failure clinic (standard care), plus a "Discharge Packet for Patients Diagnosed with Heart Failure", developed by the American Heart Association. Both groups will be asked via text messages and/or telephone calls to complete questionnaires at baseline/start, 4 weeks and 12 weeks, about self-care, quality of life, health beliefs, medications, diet, etc.

Participants assigned to the intervention group will also receive approximately 5 text messages/week targeting medication adherence, heart-healthy diet, and self-monitoring for 12 weeks.

DETAILED DESCRIPTION:
Heart failure (HF) is a serious chronic condition and the most common hospital discharge diagnosis among older adults in the United States. Almost 7 million Americans are diagnosed with HF and new cases are rapidly rising at a rate of nearly 1 million per year. This feasibility pilot randomized controlled trial will be conducted using individually tailored text message (TM) intervention, delivered to improve HF self-care adherence.

This randomized controlled trial in older adult patients (≥50 years of age) with HF to determine the feasibility (recruitment capability, acceptability), and preliminary efficacy of the Text4HF intervention compared with usual care over 12 weeks. Thirty (n=30) adult patients from the University of Illinois Hospital & Health Sciences System (UIH) will be randomly assigned to the intervention or usual care group. Patients in the TM intervention (TEXT4HF) will receive messages that target the most common self-care factors known to precipitate HF hospitalizations (medication adherence, heart-healthy diet, and self-monitoring).

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of Age
* HF Stage C, NYHA Class I-IV and on a loop diuretic
* Own a Mobile phone with Text message plan
* Ability to speak and read English
* Suboptimal HF self-care. (SCHFI Score of 3 or less in at least 2 items of any subscale: Self-care maintenance, Symptom Perception, or Self-management)

Exclusion Criteria:

* SAVR/TAVR or Ventricular Assist Device, or Cardiac Resynchronization Therapy (CRT) - implantation, and/or heart transplantation (HTx) scheduled within the next 3 months
* Coronary revascularization, and/or CRT-implantation within the last 30 days (EMR Review)
* Psychosis
* Hospice or End-of-life care
* Advanced Renal disease (i.e., estimated Glomerular Filtration Rate <25 or Hemodialysis)
* Cognitive impairment (i.e., Dementia, Alzheimer's)
* Unable to self-manage (take medication, bathe, use the toilet, etc.)
* Currently living in a nursing home

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Care Maintenance | Baseline, 4 weeks, 12 weeks
  Self-care maintenance will be measured with Subscale A of the Self-Care Heart Failure Index (SCHFI) v.7.2, which includes 10-items. Standardized scores in this scale range from 0 to 100. A total score of ≥70 indicates adequate self-care.
Change in Self-care Symptom Perception | Baseline, 4 weeks, 12 weeks
  Self-care symptom perception will be measured the Self-Care Heart Failure Index (SCHFI) v.7.2, Subscale B, which includes 9-items. Standardized scores in this scale range from 0 to 100. A total score of ≥70 indicates adequate self-care.
Change in Self-care self-management | Baseline, 4 weeks, 12 weeks
  Self-care self-management will be measured with the Self-Care Heart Failure Index (SCHFI) v.7.2, Subscale C, which includes 8-items. Standardized scores in this scale range from 0 to 100. A total score of ≥70 indicates adequate self-care.

SECONDARY OUTCOMES:
Health Beliefs about Medication Compliance | Baseline, 4 weeks, 12 weeks
  Beliefs about Medication Compliance Scale (12-items)The instrument uses a 5-point Likert scale. Benefits and Barriers scores range from 6-30. Lower Barrier scores indicate a better outcome. Higher Benefits scores indicate a better outcome.
Health Beliefs about Dietary Compliance | Baseline, 4 weeks, 12 weeks
  Beliefs about Dietary Compliance Scale (12 items)The instrument uses a 5-point Likert scale. Benefits and Barriers scores range from 6-30. Lower Barrier scores indicate a better outcome. Higher Benefits scores indicate a better outcome.
Health Beliefs about Self-Monitoring Compliance | Baseline, 4 weeks, 12 weeks
  Beliefs about Self-Monitoring Scale (18 items). The instrument uses a 5-point Likert scale. Benefits and Barriers scores range from 18-90. Lower Barrier scores indicate a better outcome. Higher Benefits scores indicate a better outcome.
Heart Failure knowledge | Baseline, 4 weeks, 12 weeks
  Atlanta Heart Failure Knowledge Questionnaire (30-items). Scored range is 0 to 30 with higher scored indicating better knowledge about heart failure.
Change in Self-care confidence (self-efficacy) | Baseline, 4 weeks, 12 weeks
  Self-care confidence ill be measured with the Self-Care Heart Failure Index (SCHFI) v.7.2, Subscale D, which includes 10-items. Standardized scores in this scale range from 0 to 100. A total score of ≥70 indicates adequate self-care.
Medication and Refill adherence | Baseline, 4 weeks, 12 weeks
  Assessed with Adherence to Refilling Medication Scale (ARMS); 12 Items, 4-point Likert scale, lower scores indicate better adherence
Heart Healthy Diet Adherence | Baseline, 4 weeks, 12 weeks
  Assessed with Scale for Dietary Behaviors in Heart Failure (SDBHF); 19 Items, 4-point Likert scale, higher scores indicate better adherence
Heart Failure Quality of Life | Baseline, 4 weeks, 12 weeks
  Assessed with Minnesota Living with Heart Failure Questionnaire; 21 questions, 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Leigh, MPH, MSHI, Principal Investigator — University of Illinois Chicago; Spyros Kitsiou, PhD, Study Chair — University of Illinois Chicago
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No